CLINICAL TRIAL: NCT01964326
Title: A Multicenter, Actual Use Trial In A Simulated Over-the-counter Environment Of Atorvastatin Calcium 10 Mg
Brief Title: Actual Use Trial of Atorvastatin Calcium 10 mg
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Not Applicable | Masking: None | Purpose: Treatment
Other Study IDs: A2581189
Record Dates: First submitted 2013-10-14; First posted 2013-10-17 (Estimated); Results first posted 2016-01-27 (Estimated); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Hypercholesterolemia
Keywords: atorvastatin; Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Atorvastatin calcium 10 mg (Experimental)
  Interventions: Drug: Atorvastatin calcium 10 mg

INTERVENTIONS:
Drug: Atorvastatin calcium 10 mg — Atorvastatin calcium 10 mg tablet to be administered orally every day

SUMMARY:
The purpose of this actual use study is to simulate the over the counter use of atorvastatin calcium 10 mg.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age (19 in Alabama).
* Provide written informed consent.
* Never participated in a study about cholesterol medicines.

Exclusion Criteria:

* Females subjects who are pregnant or breastfeeding.
* Subjects with active liver disease.
* Subjects taking cyclosporine.
* Subjects with a known allergy to atorvastatin calcium.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1311 (Actual)
Dates: Start 2013-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (37):
- United States (37):
  - Robert's Discount Pharmacy, Hoover, Alabama
  - Pharmacy at the Pig, McCalla, Alabama
  - Pinson Discount Drugs, Pinson, Alabama
  - Community Clinical Pharmacy, Mesa, Arizona
  - Melrose Pharmacy, Phoenix, Arizona
  - Bi-Rite Quality Pharmacies, La Habra, California
  - Parkview Compounding Pharmacy, Rancho Cucamonga, California
  - Garden Drug, Fort Lauderdale, Florida
  - Pill Box Pharmacy and Medical Supply, Pembroke Pines, Florida
  - Summerfield Pharmacy, Riverview, Florida
  - Sutton Family Pharmacy, Dalton, Georgia
  - Wynn's Pharmacy Inc., Griffin, Georgia
  - Catonsville Pharmacy, Baltimore, Maryland
  - Kemper Drug, Elk River, Minnesota
  - Goodrich Pharmacy, Fridley, Minnesota
  - Northfield Pharmacy, Northfield, Minnesota
  - Cub Pharmacy, Rosemount, Minnesota
  - Goodrich Pharmacy, Saint Francis, Minnesota
  - Albers' Medical Pharmacy, Kansas City, Missouri
  - Countryside Pharmacy, Savannah, Missouri
  - Texas Road Pharmacy, Monroe, New Jersey
  - Duran Central Pharmacy, Albuquerque, New Mexico
  - Sam's Regent Pharmacy, Albuquerque, New Mexico
  - Family Prescription Center, Bethlehem, Pennsylvania
  - T.B. Bond Pharmacy, Hillsboro, Texas
  - Inwood Pharmacy, Houston, Texas
  - Brick Street Pharmacy, Tyler, Texas
  - Mountain West Apothecary, Bountiful, Utah
  - Ridgeview Pharmacy, Roy, Utah
  - The Apothecary Shoppe, Salt Lake City, Utah
  - The Medicine Center, Salt Lake City, Utah
  - Family Plaza Pharmacy, West Jordan, Utah
  - Montpelier Pharmacy, Inc., Montpelier, Virginia
  - Lafayette Pharmacy, Richmond, Virginia
  - Jim's Pharmacy, Enumclaw, Washington
  - Ostrom Drugs, Kenmore, Washington
  - Katterman's Sand Point Professional Pharmacy, Seattle, Washington

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A2581189&StudyName=Actual%20Use%20Trial%20of%20Atorvastatin%20Calcium%2010%20mg%20

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were screened by phone, then referred to their participating retail pharmacy site for a scheduled face-to-face interview, after which they were given an empty atorvastatin(Lipitor) over-the-counter(OTC) package to review the information on the outside of the entire package,after which decision was made to purchase the medicine by them.
Groups:
- Atorvastatin: Participants after reading the drugs fact label (DFL), made a purchase decision, purchased (on Day 1) and used atorvastatin 10 milligram (mg) OTC for 26 weeks.
Period: Overall Study
Arm/Group | Atorvastatin
Started | 1311
Completed | 1014
Not Completed | 297
Not completed — Adverse Event | 48
Not completed — Death | 2
Not completed — Protocol Violation | 4
Not completed — Lost to Follow-up | 88
Not completed — Withdrawal by Subject | 87
Not completed — Pregnancy | 1
Not completed — No Longer Meets Eligibility Criteria | 1
Not completed — Physician Decision | 55
Not completed — Investigator Discretion | 1
Not completed — Other | 9
Not completed — Did not meet eligibility criteria | 1

BASELINE CHARACTERISTICS:
Population: Users/Safety set included all participants reported taking at least 1 dose of study medication or had at least 1 dosing record available or responded 'yes' to the question 'have you started taking Lipitor OTC' in any phone interview, or contacted the study site in any other manner and indicated the use of study product.
Arm/Group | Atorvastatin
Number analyzed (Participants) | 1234
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.8 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 593
  Male | 641

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Complied With the Direction to Check Their Low-density Lipoprotein Cholesterol (LDL-C) Level
Description: Percentage of participants whose behavior was either correct or acceptable were considered to be compliant. The behavior was considered correct if participants had their LDL-C checked between Weeks 4 and 12. The behavior was considered acceptable if participants had their LDL-C checked between Weeks 2 and 3 (before Week 4) or between Weeks 13 (after Week 12) and 26 or if participants were instructed by a physician that an LDL-C test was not needed.
Time Frame: Day 1 up to Week 26
Population: The analysis was performed on the continuing users set which is a subset of the users set, defined as the users who continued taking the study medication for at least 6 weeks since the first date of the study treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Atorvastatin
Number analyzed (Participants) | 1041
Percentage of participants | 49.7 [46.6 to 52.7]

2. Primary Outcome: Percentage of Participants Who Took Appropriate Action Based on Their LDL-C Results
Description: Percentage of participants whose behavior was either correct or acceptable were considered to be compliant. The behavior was considered correct if participants self-reported an LDL-C level below 130 milligram per deciliter (mg/dL) or normal, or low and decided to continue with atorvastatin OTC or if participants self-reported an LDL-C below 130 mg/dL, or normal, or low but stopped the use because of new conditions preventing them from continuing use. The behavior was considered acceptable if participants self-report LDL-C level between 130 and 135 mg/dL and continued to use atorvastatin OTC without contacting a physician or other health care practitioner or if participants self-reported LDL-C greater than or equal to (>=) 130 mg/dL('borderline high' or 'high' LDL-C), and contacted a physician after getting the LDL-C test results.
Time Frame: Day 1 up to Week 26
Population: The analysis was performed on continuing users who checked their LDL-C during the study.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Atorvastatin
Number analyzed (Participants) | 542
Percentage of participants | 52.6 [48.4 to 56.8]

3. Secondary Outcome: Percentage of Participants Taking an "Ask a Doctor or Pharmacist Before Use" Medication Who Followed the Labeling and Contacted a Doctor or Pharmacist Before Using Study Medication
Description: Percentage of participants whose behavior was either correct or acceptable were considered to be compliant. 'Ask a doctor or pharmacist before use' medication included human immunodeficiency virus (HIV) medicine, digoxin, telaprevir, rifampin, colchicine, or oral contraceptives. The behavior of the participants was considered correct if participants asked a doctor or pharmacist before use. The behavior was considered acceptable if participants contacted a doctor or pharmacist within 7 days of initiating therapy.
Time Frame: Day 1 up to Week 26
Population: The analysis was performed on the participants from the user set who reported the use of any "Ask a doctor or pharmacist before use" medication.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Atorvastatin
Number analyzed (Participants) | 24
Percentage of participants | 29.2 [11.0 to 47.4]

4. Secondary Outcome: Percentage of Participants Who Stopped Study Medication Use and Asked a Doctor if They Experienced Any of the Labeled "Stop Use and Ask a Doctor" Symptoms
Description: Percentage of participants whose behavior was either correct or acceptable were considered to be compliant. The "Stop use and ask a doctor" symptoms included: (a) unexplained muscle pain or weakness or tenderness, (b) unusual fatigue, (c) loss of appetite (d) upper belly pain (e) dark-colored urine or (f) yellowing of the whites of eyes or skin. The behavior of the participants was considered correct if participants stopped use and contacted a doctor within 7 days after the event (symptom development).The behavior was considered acceptable if participants either stopped use or contacted a doctor (but did not do both) within the 7 days' timeframe.
Time Frame: Day 1 up to Week 26
Population: The analysis was performed on the participants from the user set who experienced any of the labeled "Stop use and ask a doctor" symptoms.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Atorvastatin
Number analyzed (Participants) | 118
Percentage of participants | 10.2 [4.7 to 15.6]

ADVERSE EVENTS:
Time Frame: Day 1 up to Week 26
Description: Analysis was performed in the safety population defined as all participants who purchased the product and provided any exposure data.
Arm/Group | Atorvastatin
Serious Adverse Events (participants affected / at risk) | 53/1234
Other Adverse Events (participants affected / at risk) | 589/1234
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Atorvastatin (N=1234)
Anaemia (Blood and lymphatic system disorders) | 2
Coronary artery disease (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Coronary artery occlusion (Cardiac disorders) | 1
Goitre (Endocrine disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Chest pain (General disorders) | 1
Death (General disorders) | 2
Hernia (General disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 2
Gallbladder perforation (Hepatobiliary disorders) | 1
Bronchitis (Infections and infestations) | 2
Appendicitis (Infections and infestations) | 1
Clostridium difficile colitis (Infections and infestations) | 1
Kidney infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Septic arthritis staphylococcal (Infections and infestations) | 1
Lung abscess (Infections and infestations) | 1
Osteomyelitis (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Ankle fracture (Injury, poisoning and procedural complications) | 2
Skin abrasion (Injury, poisoning and procedural complications) | 1
Concussion (Injury, poisoning and procedural complications) | 1
Femur fracture (Injury, poisoning and procedural complications) | 1
Multiple fractures (Injury, poisoning and procedural complications) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Syncope (Nervous system disorders) | 2
Cerebrovascular accident (Nervous system disorders) | 3
Carotid artery disease (Nervous system disorders) | 1
Generalised tonic-clonic seizure (Nervous system disorders) | 1
Depression (Psychiatric disorders) | 2
Suicidal ideation (Psychiatric disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 2
Calculus bladder (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Vocal cord disorder (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Atorvastatin (N=1234)
Anaemia (Blood and lymphatic system disorders) | 3
Lymphadenopathy (Blood and lymphatic system disorders) | 2
Cardiac failure congestive (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 1
Vertigo (Ear and labyrinth disorders) | 5
Ear pain (Ear and labyrinth disorders) | 2
Tinnitus (Ear and labyrinth disorders) | 2
Hypothyroidism (Endocrine disorders) | 2
Vision blurred (Eye disorders) | 2
Conjunctivitis (Eye disorders) | 1
Eye haemorrhage (Eye disorders) | 1
Eye irritation (Eye disorders) | 1
Eyelid irritation (Eye disorders) | 1
Ocular hyperaemia (Eye disorders) | 1
Ocular icterus (Eye disorders) | 1
Optic nerve disorder (Eye disorders) | 1
Visual acuity reduced (Eye disorders) | 1
Vitreous detachment (Eye disorders) | 1
Vitreous floaters (Eye disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 40
Nausea (Gastrointestinal disorders) | 26
Constipation (Gastrointestinal disorders) | 17
Abdominal pain upper (Gastrointestinal disorders) | 16
Vomiting (Gastrointestinal disorders) | 11
Abdominal discomfort (Gastrointestinal disorders) | 9
Abdominal pain (Gastrointestinal disorders) | 8
Flatulence (Gastrointestinal disorders) | 8
Dry mouth (Gastrointestinal disorders) | 6
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 6
Toothache (Gastrointestinal disorders) | 5
Abdominal distension (Gastrointestinal disorders) | 4
Dysgeusia (Gastrointestinal disorders) | 4
Dyspepsia (Gastrointestinal disorders) | 4
Haemorrhoids (Gastrointestinal disorders) | 3
Colitis (Gastrointestinal disorders) | 2
Food poisoning (Gastrointestinal disorders) | 2
Breath odour (Gastrointestinal disorders) | 1
Faeces discoloured (Gastrointestinal disorders) | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 1
Glossitis (Gastrointestinal disorders) | 1
Glossodynia (Gastrointestinal disorders) | 1
Haematochezia (Gastrointestinal disorders) | 1
Lip dry (Gastrointestinal disorders) | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1
Swollen tongue (Gastrointestinal disorders) | 1
Tongue discolouration (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 23
Peripheral swelling (General disorders) | 9
Chest pain (General disorders) | 7
Pain (General disorders) | 4
Swelling (General disorders) | 4
Asthenia (General disorders) | 2
Tenderness (General disorders) | 2
Thirst (General disorders) | 2
Calcinosis (General disorders) | 1
Chest discomfort (General disorders) | 1
Chills (General disorders) | 1
Cyst (General disorders) | 1
Feeling abnormal (General disorders) | 1
Feeling jittery (General disorders) | 1
Influenza like illness (General disorders) | 1
Mass (General disorders) | 1
Pyrexia (General disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Gallbladder pain (Hepatobiliary disorders) | 1
Hepatitis (Hepatobiliary disorders) | 1
Seasonal allergy (Immune system disorders) | 6
Dermatitis allergic (Immune system disorders) | 1
Hypersensitivity (Immune system disorders) | 1
Nasopharyngitis (Infections and infestations) | 44
Influenza (Infections and infestations) | 19
Sinusitis (Infections and infestations) | 18
Urinary tract infection (Infections and infestations) | 17
Bronchitis (Infections and infestations) | 15
Pneumonia (Infections and infestations) | 5
Upper respiratory tract infection (Infections and infestations) | 4
Gastroenteritis (Infections and infestations) | 3
Herpes zoster (Infections and infestations) | 3
Skin infection (Infections and infestations) | 3
Viral infection (Infections and infestations) | 3
Fungal infection (Infections and infestations) | 2
Labyrinthitis (Infections and infestations) | 2
Respiratory tract infection (Infections and infestations) | 2
Tooth abscess (Infections and infestations) | 2
Tooth infection (Infections and infestations) | 2
Vaginal infection (Infections and infestations) | 2
Acarodermatitis (Infections and infestations) | 1
Bacterial vaginosis (Infections and infestations) | 1
Bursitis infective (Infections and infestations) | 1
Candida infection (Infections and infestations) | 1
Cestode infection (Infections and infestations) | 1
Clostridium difficile colitis (Infections and infestations) | 1
Diverticulitis (Infections and infestations) | 1
Ear infection (Infections and infestations) | 1
Folliculitis (Infections and infestations) | 1
Gastric infection (Infections and infestations) | 1
Genital herpes (Infections and infestations) | 1
Hepatitis B (Infections and infestations) | 1
Infected cyst (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Kidney infection (Infections and infestations) | 1
Localised infection (Infections and infestations) | 1
Otitis media (Infections and infestations) | 1
Skin bacterial infection (Infections and infestations) | 1
Wound infection (Infections and infestations) | 1
Procedural pain (Injury, poisoning and procedural complications) | 9
Ligament sprain (Injury, poisoning and procedural complications) | 8
Muscle strain (Injury, poisoning and procedural complications) | 7
Contusion (Injury, poisoning and procedural complications) | 4
Arthropod bite (Injury, poisoning and procedural complications) | 3
Concussion (Injury, poisoning and procedural complications) | 2
Tendon injury (Injury, poisoning and procedural complications) | 2
Ankle fracture (Injury, poisoning and procedural complications) | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 1
Exposure during pregnancy (Injury, poisoning and procedural complications) | 1
Foot fracture (Injury, poisoning and procedural complications) | 1
Foreign body in eye (Injury, poisoning and procedural complications) | 1
Hand fracture (Injury, poisoning and procedural complications) | 1
Injury (Injury, poisoning and procedural complications) | 1
Injury corneal (Injury, poisoning and procedural complications) | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1
Laceration (Injury, poisoning and procedural complications) | 1
Limb crushing injury (Injury, poisoning and procedural complications) | 1
Limb injury (Injury, poisoning and procedural complications) | 1
Meniscus injury (Injury, poisoning and procedural complications) | 1
Nail injury (Injury, poisoning and procedural complications) | 1
Rotator cuff syndrome (Injury, poisoning and procedural complications) | 1
Splinter (Injury, poisoning and procedural complications) | 1
Stress fracture (Injury, poisoning and procedural complications) | 1
Wound (Injury, poisoning and procedural complications) | 1
Blood pressure increased (Investigations) | 9
Blood glucose increased (Investigations) | 8
Weight increased (Investigations) | 8
Blood cholesterol increased (Investigations) | 5
Hepatic enzyme increased (Investigations) | 3
Heart rate increased (Investigations) | 2
Liver function test abnormal (Investigations) | 2
Blood pressure decreased (Investigations) | 1
Blood urine present (Investigations) | 1
Heart rate irregular (Investigations) | 1
Platelet count increased (Investigations) | 1
Prostate examination abnormal (Investigations) | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 5
Dehydration (Metabolism and nutrition disorders) | 4
Decreased appetite (Metabolism and nutrition disorders) | 2
Fluid retention (Metabolism and nutrition disorders) | 2
Glucose tolerance impaired (Metabolism and nutrition disorders) | 2
Increased appetite (Metabolism and nutrition disorders) | 2
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 53
Arthralgia (Musculoskeletal and connective tissue disorders) | 26
Pain in extremity (Musculoskeletal and connective tissue disorders) | 20
Muscle spasms (Musculoskeletal and connective tissue disorders) | 18
Back pain (Musculoskeletal and connective tissue disorders) | 12
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 10
Arthritis (Musculoskeletal and connective tissue disorders) | 9
Gout (Musculoskeletal and connective tissue disorders) | 7
Muscular weakness (Musculoskeletal and connective tissue disorders) | 7
Joint stiffness (Musculoskeletal and connective tissue disorders) | 3
Joint swelling (Musculoskeletal and connective tissue disorders) | 3
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2
Arthropathy (Musculoskeletal and connective tissue disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 1
Diastasis recti abdominis (Musculoskeletal and connective tissue disorders) | 1
Epicondylitis (Musculoskeletal and connective tissue disorders) | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1
Synovitis (Musculoskeletal and connective tissue disorders) | 1
Tendon discomfort (Musculoskeletal and connective tissue disorders) | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 1
Trigger finger (Musculoskeletal and connective tissue disorders) | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Thyroid cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Headache (Nervous system disorders) | 37
Dizziness (Nervous system disorders) | 14
Migraine (Nervous system disorders) | 5
Hypoaesthesia (Nervous system disorders) | 4
Memory impairment (Nervous system disorders) | 4
Sciatica (Nervous system disorders) | 4
Burning sensation (Nervous system disorders) | 2
Convulsion (Nervous system disorders) | 2
Neuralgia (Nervous system disorders) | 2
Paraesthesia (Nervous system disorders) | 2
Anal sphincter atony (Nervous system disorders) | 1
Disorientation (Nervous system disorders) | 1
Disturbance in attention (Nervous system disorders) | 1
Muscular weakness (Nervous system disorders) | 1
Paraesthesia oral (Nervous system disorders) | 1
Restless legs syndrome (Nervous system disorders) | 1
Stupor (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 8
Insomnia (Psychiatric disorders) | 8
Depression (Psychiatric disorders) | 6
Confusional state (Psychiatric disorders) | 2
Nervousness (Psychiatric disorders) | 2
Nightmare (Psychiatric disorders) | 2
Affect lability (Psychiatric disorders) | 1
Panic attack (Psychiatric disorders) | 1
Sleep disorder (Psychiatric disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 6
Chromaturia (Renal and urinary disorders) | 4
Bladder pain (Renal and urinary disorders) | 1
Pollakiuria (Renal and urinary disorders) | 1
Urine odour abnormal (Renal and urinary disorders) | 1
Erectile dysfunction (Reproductive system and breast disorders) | 4
Breast abscess (Reproductive system and breast disorders) | 1
Breast mass (Reproductive system and breast disorders) | 1
Libido decreased (Reproductive system and breast disorders) | 1
Menorrhagia (Reproductive system and breast disorders) | 1
Ovarian cyst (Reproductive system and breast disorders) | 1
Spontaneous penile erection (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 10
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 2
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1
Nasal disorder (Respiratory, thoracic and mediastinal disorders) | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 11
Pruritus (Skin and subcutaneous tissue disorders) | 6
Skin lesion (Skin and subcutaneous tissue disorders) | 3
Swelling face (Skin and subcutaneous tissue disorders) | 2
Acne (Skin and subcutaneous tissue disorders) | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Eczema (Skin and subcutaneous tissue disorders) | 1
Ingrown hair (Skin and subcutaneous tissue disorders) | 1
Lichen planus (Skin and subcutaneous tissue disorders) | 1
Onychoclasis (Skin and subcutaneous tissue disorders) | 1
Rash generalised (Skin and subcutaneous tissue disorders) | 1
Rash papular (Skin and subcutaneous tissue disorders) | 1
Skin disorder (Skin and subcutaneous tissue disorders) | 1
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Victim of sexual abuse (Social circumstances) | 1
Flushing (Vascular disorders) | 2
Hypertension (Vascular disorders) | 2
Hypotension (Vascular disorders) | 2
Thrombosis (Vascular disorders) | 2
Arteriosclerosis (Vascular disorders) | 1
Haematoma (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.